CLINICAL TRIAL: NCT00149708
Title: Consequence of Lifetime Isolated Growth Hormone Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: roberto salvatori, MD, Johns Hopkins University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK 65718 (completed)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth hormone; Deficiency; Cardiovascular risk; Body composition
MeSH Terms: conditions — Dwarfism, Pituitary

INTERVENTIONS:
Drug: growth hormone administration for 6 months — depot GH (Nutropin depot) 13.4 mg every 14 days
  Other Names: Nuropin depot

SUMMARY:
Growth hormone (GH) deficiency (GHD) in adulthood has been associated with changes in body composition (e.g. increased abdominal obesity, and reduced muscle mass), in organ functions (e.g. reduced cardiac systolic function), in metabolic parameters linked to increased risk of cardiovascular disease (e.g. increased serum total and LDL cholesterol, C reactive protein, and plasma fibrinogen), and with reduced bone density. These observations have been used to define the "adult GHD syndrome" and to advocate GH replacement therapy in GHD adults. However, most of the studies have been performed in patients who have had hypothalamic or pituitary diseases, and/or have undergone brain irradiation. Such patients are often chronically sick, and commonly lack other pituitary hormones, whose replacement therapies may not fully restore the physiological functions of the under-active glands. Reliable data on the existence of the AGHD syndrome and its response to GH therapy can be only obtained by studying patients that are otherwise healthy. However, isolated GH deficiency (IGHD) is a rare disease. In addition, up to 50% of patients who have been diagnosed with IGHD in childhood are no longer GH deficient as adults, making such study difficult to perform due to the scarcity of patients population. We have identified a very large homogeneous population of patients who have IGHD due to a homozygous mutation in the GHRH-receptor (GHRHR) gene that resides in a rural area of Brazil. None of the adult dwarf patients has ever been treated with hGH replacement. This population represents a unique model to study the effect of isolated lifetime lack of GH. We propose studies of physiological and metabolic parameters in subjects who are homozygous for this mutation and compare them with normal subjects residing in the same community.

The primary goal of this proposal is to determine the consequences of life-long lack of GH on body composition, muscle strength, cardiovascular status, cardiovascular risk factors, thyroid status and bone density and metabolism, and to test which of these parameters are reversed by a 6-month course of GH replacement therapy. In addition, we want to test the hypothesis that heterozygosity for this GHRHR mutation causes a phenotype that may be intermediate between the one present in homozygous normal subjects and in homozygous affected GHD patients. This is relevant because inactivating mutations in the GHRHR are being described with increasing frequency in populations of different genetic background, suggesting that individuals with faulty single GHRHR alleles may be present in significant numbers in the general population.

DETAILED DESCRIPTION:
SPECIFIC AIM 1: To study anthropometric parameters, cardiovascular and metabolic status and cardiovascular risk profile, including inflammatory markers of cardiovascular relevance, muscle strength, bone density and bone metabolism, and thyroid status of twenty GH-naïve adult GHD subjects who are homozygous for a null GHRHR mutation and to compare them with twenty age- and sex- matched normal controls from the same population.

SPECIFIC AIM 2: To observe the changes in all the above parameters that occur in GHD subjects after a 6-months treatment with hGH replacement, and their reversibility after a 6-months washout period.

SPECIFIC AIM 3: To determine effect of heterozygosity for the GHRHR mutation. To this end, we propose to genotype a large number of apparently normal members of the Itabaianinha community with the goal of separating subjects homozygous for the wild-type allele from subjects heterozygous for the GHRHR mutation, and to compare their phenotype with the one observed in subjects homozygous for the wild type allele residing in the same geographical area.

Together, these studies will determine the effect of lifetime absence of GH on multiple organ functions and their response to hGH therapy, and will tell if heterozygosity for mutations in the GHRHR gene is associated with a detectable phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Lifetime isolated and untreated growth hormone deficiency

Exclusion Criteria:

* Age below 18 years, pregnancy, diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Body composition | after 6 months of GH and after wash out (6 and 12 months)
Lipid levels | after 6 months of GH and after 6 and 12 months of wash out
Heart function | after 6 months of GH and after 6 and 12 months of wash out

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Salvatori, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Federal University of Sergipe, Aracaju, Sergipe, Brazil

REFERENCES:
- [Result] Alcantara MR, Salvatori R, Alcantara PR, Nobrega LM, Campos VS, Oliveira EC, Oliveira MH, Souza AH, Aguiar-Oliveira MH. Thyroid morphology and function in adults with untreated isolated growth hormone deficiency. J Clin Endocrinol Metab. 2006 Mar;91(3):860-4. doi: 10.1210/jc.2005-2555. Epub 2006 Jan 4. PMID 16394080
- [Derived] Araujo VP, Aguiar-Oliveira MH, Oliveira JL, Rocha HM, Oliveira CR, Rodrigues TM, Nunes MA, Britto IM, Ximenes R, Barreto-Filho JA, Meneguz-Moreno RA, Pereira RM, Valenca EH, Oliveira-Neto LA, Vicente TA, Blackford A, Salvatori R. Arrest of atherosclerosis progression after interruption of GH replacement in adults with congenital isolated GH deficiency. Eur J Endocrinol. 2012 Jun;166(6):977-82. doi: 10.1530/EJE-12-0062. Epub 2012 Mar 13. PMID 22416078
- [Derived] Barbosa JA, Salvatori R, Oliveira CR, Pereira RM, Farias CT, Britto AV, Farias NT, Blackford A, Aguiar-Oliveira MH. Quality of life in congenital, untreated, lifetime isolated growth hormone deficiency. Psychoneuroendocrinology. 2009 Jul;34(6):894-900. doi: 10.1016/j.psyneuen.2009.01.001. Epub 2009 Jan 31. PMID 19181452
- [Derived] Menezes Oliveira JL, Marques-Santos C, Barreto-Filho JA, Ximenes Filho R, de Oliveira Britto AV, Oliveira Souza AH, Prado CM, Pereira Oliveira CR, Pereira RM, Ribeiro Vicente Tde A, Farias CT, Aguiar-Oliveira MH, Salvatori R. Lack of evidence of premature atherosclerosis in untreated severe isolated growth hormone (GH) deficiency due to a GH-releasing hormone receptor mutation. J Clin Endocrinol Metab. 2006 Jun;91(6):2093-9. doi: 10.1210/jc.2005-2571. Epub 2006 Mar 7. PMID 16522693